CLINICAL TRIAL: NCT01744405
Title: Study Of Nifurtimox Transfer Into Breastmilk In Lactating Women With Chagas Disease
Acronym: LACTNFX
Status: Completed | Type: Observational
Sponsor: Hospital de Niños R. Gutierrez de Buenos Aires (Other)
Responsible Party: Principal Investigator, Facundo Garcia-Bournissen, Associate Resesarcher, Hospital de Niños R. Gutierrez de Buenos Aires
Other Study IDs: LACT-NIFURTIMOX
Record Dates: First submitted 2012-12-05; First posted 2012-12-06 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2015-03

CONDITIONS: Chagas Disease; Lactation
Keywords: Chagas disease; lactation; breastmilk; postpartum period; infants; pediatric clinical pharmacology; developmental clinical pharmacology; parasitology; trypanosoma cruzi; nifurtimox
MeSH Terms: conditions — Chagas Disease; Breast Feeding

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — breastmilk; plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Lactating Women with Chagas disease: Women with Chagas disease who fulfill clinical criteria for treatment with nifurtimox, and who are also lactating

SUMMARY:
The investigators propose to study the transfer of nifurtimox into breastmilk of lactating women who receive the drug for the treatment of Chagas disease.

Breastmilk and blood samples will be obtained from these patients at pre-specified times after they take the clinically indicated medication, and the concentrations in both matrices will be compared to estimate degree of transfer. Estimation of nifurtimox transfer into breastmilk will allow the evaluation of potential degree of exposure of infants breastfed by these women to nifurtimox. This study will help clarify safety of continuing breastfeeding while receiving treatment with nifurtimox for Chagas disease.

ELIGIBILITY:
Inclusion Criteria:

* Lactating women with Chagas disease, not treated before
* Use of contraception

Exclusion Criteria:

* History of allergy to nifurtimox or its excipients
* Pregnancy
* Significant heart involvement (due to Chagas disease)
* Significant systemic diseases that could affect the interpretation of the results in the opinion of the principal investigator

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Population of young women with Chagas disease referred to our center for evaluation and treatment
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2012-12; Primary Completion 2013-12 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Nifurtimox concentration in breastmilk and in plasma | at randomly selected, pre-specified, time points during the 30 days of treatment
  Randomly obtained breastmilk samples will be obtained to both evaluate the breastmilk / plasma concentration ratio of the drug, and to develop a population pharmacokinetics model of drug transfer into breastmilk, if possible.

SECONDARY OUTCOMES:
Incidence of adverse drug reactions in women treated with nifurtimox during lactation | throughout the 30 days of treatment
  Women receiving treatment with nifurtimox while lactating, enrolled in the study will be followed according to current clinical guidelines, and monitored during the 30 days of treatment (as per Chagas disease treatment guidelines), and monthly for 3 months after treatment completion.

CONTACTS AND LOCATIONS:
Overall Officials: Facundo Garcia Bournissen, MD PhD, Principal Investigator — Buenos Aires Children´s Hospital Ricardo Gutierrez ; CONICET
Locations (1):
- Parasitology and Chagas Service, Buenos Aires Children´s Hospital Ricardo Gutierrez, Buenos Aires, Buenos Aires, Argentina

REFERENCES:
- [Derived] Moroni S, Marson ME, Moscatelli G, Mastrantonio G, Bisio M, Gonzalez N, Ballering G, Altcheh J, Garcia-Bournissen F. Negligible exposure to nifurtimox through breast milk during maternal treatment for Chagas Disease. PLoS Negl Trop Dis. 2019 Aug 15;13(8):e0007647. doi: 10.1371/journal.pntd.0007647. eCollection 2019 Aug. PMID 31415566